CLINICAL TRIAL: NCT04311710
Title: A Phase 1/2 Pharmacokinetic Multi-tumor Study of Subcutaneous Formulation of Ipilimumab Monotherapy and in Combination With Subcutaneous Nivolumab
Brief Title: A Study Evaluating the Drug Levels of Iplimumab Given Under the Skin Alone and in Combination With Nivolumab in Multiple Tumor Types
Acronym: CheckMate 76U
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA209-76U
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Tumor
Keywords: lung cancer, renal cancer, bladder cancer, skin cancer, liver cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Skin Neoplasms; Liver Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Arm A: mM, mUC, HCC (Experimental): metastatic Melanoma (mM), metastatic Urothelial Carcinoma (mUC), and advanced Heptocellular Carcinoma (HCC)
  Interventions: Drug: ipilimumab; Drug: nivolumab; Drug: ENHANZE (rHuPH20)
- Part 1: Arm B: mM (Experimental): metastatic Melanoma (mM)
  Interventions: Drug: ipilimumab; Drug: nivolumab
- Part 2: Arm A: NSCLC (Experimental): metastatic non small cell lung cancer (NSCLC)
  Interventions: Drug: ipilimumab; Drug: ENHANZE (rHuPH20); Drug: nivolumab
- Part 2: Arm B: RCC (Experimental): advanced or metastatic renal cell carcinoma (RCC)
  Interventions: Drug: ipilimumab; Drug: ENHANZE (rHuPH20); Drug: nivolumab

INTERVENTIONS:
Drug: ipilimumab — Specified Dose on Specified Days
  Other Names: (BMS-734016)
Drug: nivolumab — Specified Dose on Specified Days
  Other Names: (BMS-936558)
  Arms: Part 1 Arm A: mM, mUC, HCC; Part 1: Arm B: mM
Drug: ENHANZE (rHuPH20) — Specified Dose on Specified Days
  Arms: Part 1 Arm A: mM, mUC, HCC; Part 2: Arm A: NSCLC; Part 2: Arm B: RCC
Drug: nivolumab — Specified Dose on Specified Days
  Other Names: (BMS-986298)
  Arms: Part 2: Arm A: NSCLC; Part 2: Arm B: RCC

SUMMARY:
A study evaluating the drug levels of ipilimumab alone and in combination with nivolumab applied under the skin in various tumor types

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Men and women must follow methods of contraception as described in the protocol

Part 1 Arms A and B: Metastatic Melanoma

- Previously untreated, histologically confirmed stage IV melanoma, as per American Joint Committee on Cancer (AJCC) staging system v.8.0

Part 1 Arm A:Advanced/mUC - Participants with histologically or cytologically confirmed urothelial carcinoma.

Part 1 Arm A: Advanced HCC

* Participants with histological confirmation of Hepatocellular Cancer (HCC)

Part 2 Arm A: Metastatic NSCLC

- Participants with histologically confirmed stage IV or recurrent Non Small Cell Lung Cancer (NSCLC)

Part 2 Arm B: Advanced or Metastatic RCC

* Histological confirmation of Renal Cell Carcinoma (RCC)
* ECOG Performance Status of 0 or 1 and for RCC (Part 2 Arm B), Karnofsky performance status ≥ 70%

Exclusion Criteria:

- History of allergy or hypersensitivity to study drug components

Part 1 Arm A: Advanced HCC

* History of hepatic encephalopathy or evidence of portal hypertension
* Active coinfection with hepatitis D virus infection in participants with HBV

Part 2 Arm A:Metastatic NSCLC

- Participants with known ALK translocations and EGFR mutation that are sensitive to available targeted inhibitor therapy

Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Part 1 Arm A: Average concentration of ipilimumab (Cavg21d) | Day 21
Part 1 Arm A: Area under the concentration in ipilimumab AUC(0-21d) | Day 21
Part 1 Arm A: Maximum observed serum concentration of ipilimumab (Cmax) | Up to 21 days
Part 1 Arm A: Observed concentration of ipilimumab at 21 days post dose (C21d) | Day 21
Part 1 Arm A: Time of maximum observed concentration in ipilimumab (Tmax) | Up to 21 days
Part 2 Arm A: Average concentration in ipilimumab (Cavg42d) | Day 42
Part 2 Arm A: Area under the concentration in ipilimumab AUC(0-42d) | Day 42
Part 2 Arm A: Maximum observed serum Concentration of Ipilimumab (Cmax) | Up to 42 days
Part 2 Arm A: Observed concentration in ipilimumab (C42d) | Day 42
Part 2 Arm A: Time of maximum observed concentration in ipilimumab (Tmax) | Up to 42 days
Part 2 Arm B: Average concentration of Ipilimumab at 21 days post dose (Cavg21d) | Day 21
Part 2 Arm B: Area Under the Concentration in Ipilimumab AUC(0-21d) | Day 21
Part 2 Arm B: Maximum observed serum Concentration in Ipilimumab (Cmax) | Up to 21 days
Part 2 Arm B: Observed concentration of ipilimumab at 21 days post dose (C21d) | Day 21
Part 2 Arm B: Time of maximum observed concentration in Ipilimumab (Tmax) | Up to 21 days

SECONDARY OUTCOMES:
Part 1 Arm B: Average concentration of ipilimumab without rHuPH20 (Cavg21d) | Day 21
Part 1 Arm B: Area under the concentration in ipilimumab without rHuPH20 AUC(0-21d) | Day 21
Part 1 Arm B: Maximum observed serum concentration of ipilimumab without rHuPH20 (Cmax) | Up to 21 days
Part 1 Arm B: Observed concentration of ipilimumab without rHuPH20 at 21 days post dose (C21d) | Day 21
Part 1 Arm B: Time of maximum observed concentration in ipilimumab without rHuPH20 (Tmax) | Up to 21 days
Incidence of adverse events (AE's) | Up to 2.5 years
Incidence of serious adverse events (SAEs) | Up to 5 years
Incidence of AE's leading to discontinuation | Up to 2.5 years
Incidence of death | Up to 2.5 years
Incidence of laboratory abnormalities | Up to 2.5 years
Instance of Anaphylactic occurring within 2 days of study drug administration | Up to 2.5 years
Instance of hypersensitivity occurring within 2 days of study drug administration | Up to 2.5 years
Incidence of hypersensitivity occurring within 2 days of study drug administration | Up to 2.5 years
Incidence of infusion reactions occurring within 2 days of study drug administration | Up to 2.5 years
Incidence of injection occurring within 2 days of study drug administration | Up to 2.5 years
Percentage of participants who develop anti-ipilimumab antibodies | Up to 2.5 years
Percentage of participants who develop anti-nivolumab antibodies | Up to 2.5 years
Percentage of participants who have developed neutralizing antibodies | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (2):
  - Local Institution - 0020, Hartford, Connecticut
  - Local Institution - 0013, Fort Wayne, Indiana
- Italy (3):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-s.c. melanoma, immunoterapia oncologica e terapie, Napoli
  - Humanitas-U.O di Oncologia medica ed Ematologia, Rozzano
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica, Siena
- Local Institution - 0010, Auckland, New Zealand

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm